CLINICAL TRIAL: NCT03541070
Title: The Effect of Kinesiology Taping on Balance in Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güllü AYDIN, Research Assistant Güllü AYDIN, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KA-17070-1
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Balance; Duchenne Muscular Dystrophy
Keywords: kinesiology taping; balance; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kinesiology taping (Experimental): For tibialis anterior muscle taping, each children's feet were placed at plantar flexion and eversion position while knees were extended, and I-shaped band was applied over tibialis anterior from origin to insertion of muscle with approximately 25-50% tension of the original length of the band. No tension was applied to the first and last 5 cm section of the bands in both applications because it were used as anchor. The tapes were remained for 1 hour on skin of both quadriceps and tibialis anterior muscles, and in this time the children were rested.
  Interventions: Device: Kinesiology tape

INTERVENTIONS:
Device: Kinesiology tape — Kinesiology taping (KT) was developed by Kenzo Kase in the 1970s. KT has similar thickness and flexibility to the skin. These tapes are used in orthopedic and sports injuries as well as neurological and rheumatic diseases, pediatric patients, lymph edema and painful conditions. These tapes are used for correcting muscle function, increasing circulation, increasing proprioception, reducing pain, and repositioning the sublease joint according to the usage method

SUMMARY:
Investigators investigated that the effects of kinesilogy taping on balance in patients with Duchenne Muscular Dystrophy

DETAILED DESCRIPTION:
Forty-five patients from Level 1 and 2 according to the Brooke Lower Extremity Functional Classification were included in the study. Balance was assessed by Pediatric Berg Balance Test (PBBT), Timed and Go Test (TUGT), and standing on one leg test. Kinesiology taping (KT) with facilitation technique was applied on bilateral quadriceps and tibialis anterior muscles and the assessments were repeated 1 hour after application. The comparison between before and after taping was analyzed.

ELIGIBILITY:
Inclusion Criteria:

DMD diagnosis being Level I and II according to Brooke Lower Extremity Functional Classification no cooperation problem no injury or orthopedic/neurologic surgery within the past 6 months no severe contracture at ankle

Exclusion Criteria:

children who did not meet the above criteria were not included

Ages: 5 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Balance Test-Timed up and go test | About 15 seconds
  Timed up and go test is a valid and practical objective measure for the pediatric population that measuring various components such as walking speed, postural control, functional mobility and balance. The children were asked to stand up from a chair, walk during 3 meters, turn, and walk back to chair and sit down. This time was recorded as second

SECONDARY OUTCOMES:
Pediatric Berg Balance Test | 15 minutes
  Pediatric Berg Balance Test is a modified version of the Berg Balance Scale that a valid and reliable test for the elderly population, for children in school age with mild to moderate motor impairment. The patients were asked to maintain their balance at the positions indicated in the test. The score of each item varies according to the parameters of the test. The score of this test is between 0-4 and the highest total score is 56.
duration in standing on one leg | about 1 minute
  Duration in standing on right and left leg was recorded as second

CONTACTS AND LOCATIONS:
Overall Officials: Güllü Aydın, R.A, Principal Investigator — Hacettepe University; İpek Alemdaroğlu Gürbüz, Assoc. Prof., Principal Investigator — Hacettepe University; Öznur Yılmaz, Prof., Principal Investigator — Hacettepe University; Ayşe Karaduman, Prof., Principal Investigator — Hacettepe University; Numan Bulut, R.A, Principal Investigator — Hacettepe University; Haluk Topaloğlu, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)